CLINICAL TRIAL: NCT03040869
Title: Risk Factors Investigation in Young Patients With Coronary Artery Disease and Their Clinical Follow-up
Brief Title: Risk Facotors in Young CHD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xu Lei, Doctor, Shanghai Zhongshan Hospital
Other Study IDs: 2016-02-25-1
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Risk Factor, Cardiovascular, Young CHD Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHD Patients: coronary angioplasty confirmed coronary heart disease.
- non-CHD patients: coronary angioplasty confirmed no coronary heart disease.

INTERVENTIONS:
Other:

SUMMARY:
Coronary heart disease (CHD) is the leading global cause of human death. Over the past decade, level of overall diagnosis and treatment of CHD has been greatly improved due to the progression of clinical research and development of technical means and the mortality of CHD has decreased by nearly 50% in western countries [1]. However, there are surveys shows that with the improvement of living standards and changes in lifestyle, the incidence of CHD is still rising in China and other developing countries, and the prevalence trend is obvious younger [2]. The so-called young CHD, generally refers to the age at onset of CHD is less than or equal to 45 years. Compared with other age-group CHD, young CHD has the following characteristics: 1. Genetic factors have a stronger effect at younger onset ages, and incidence with obvious familial aggregation[3]; 2 Often with the onset of acute coronary syndrome, presumably may be associated with strong inflammation of the lesion; 3. Two extremes often exists in coronary lesions: mild or no atherosclerosis and severe triple-vessel disease; 4 Rapid progression of atherosclerotic lesions, stent restenosis in the same site repeated after interventional treatment, rapid progress of lesion in non-intervention site;5 Surgical mortality is low in regardless of interventional therapy or bypass surgery, but the rate of revascularization is significantly higher in following 10 years.

DETAILED DESCRIPTION:
Study method

* Recruited the patients meet the inclusion criteria since March 2016, collected the information of the change of risk factors, angina in pre-operation, mode of onset, characteristics of coronary artery, morbility of treatment,clinical follow-up; ② Collect the following information in clinical cases: gender, age, history of hypertension, history of diabetes, cholesterol level, triglyceride level, sedentary, body index, family history of CHD, genotype of ALDH2 and MTHFR, history of myocardial infarction, coronary artery lesions and operation situation; ③ The follow-up was performed through clinic and telephone every half or one year. The details include whether recurrence of angina, the main symptom, the cause of attack, lasting time, the efficacy of taking nitroglycerin, whether performed electrocardiography examination, whether occurred myocardial infarction and the attack site. whether performed interventional therapy and CABG surgery again and the cause of surgery, whether re-examined coronary arteriongraphy, whether death and the cause, and the occurred date in above events; ④ Analysis the pathogenic intensity with each risk factors with other age group CHD.

3.2 Study population 3.2.1 inclusion criteria

Young CHD group:

* Below or equal to 45 years of age;

  ② Patients suffered stable or latent coronary heart disease, unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction diagnosed by coronary angiography or coronary CT scan;

  ③ Signed informed consent form. Non-young CHD group
* Below or equal to 45 years of age;

  ② Patients suffered stable or latent coronary heart disease, unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction diagnosed by Coronary angiography or coronary CT scan;

  ③ Risk factors such as the gender, high cholesterol, high blood pressure, overweight, diabetes, smoking, homocysteine levels matched with inclusion criteria 1 subjects enrolled.

  ④ Signed informed consent form Young non-coronary heart disease
* Below or equal to 45 years of age; ② Patients were confirmed to rule out the stable or latent coronary heart disease, unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction diagnosed by Coronary angiography or coronary CT scan;

  ③ Signed Informed consent form. 3.2.2 Exclusion criteria Exclusion criteria in each group are as follows
* Patients who suffered serious liver and kidney diseases, infections, severe systemic disease such as blood disease and malignant tumor;

  ② Pregnancy or breast-feeding women;
  * Patients who could not timely follow up or refuse to participate in this study. 3.2.3 Exit criteria Subjects were claimed to withdraw informed consent. 3.3 Grouping method and cases number
* Experimental group：1250 samples

  * Positive control group：1250 samples ③ Negative control group：500 samples

ELIGIBILITY:
Inclusion Criteria:①Below or equal to 45 years of age;

②Patients suffered stable or latent coronary heart disease, unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction diagnosed by coronary angiography or coronary CT scan

Exclusion Criteria:

* Patients who suffered serious liver and kidney diseases, infections, severe systemic disease such as blood disease and malignant tumor; ②Pregnancy or breast-feeding women; ③Patients who could not timely follow up or refuse to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ①Below or equal to 45 years of age;
  ②Patients suffered stable or latent coronary heart disease, unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction diagnosed by coronary angiography or coronary CT scan;
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
heart failure | 12 months
  LVEF less than 40%

IPD SHARING:
Plan to Share IPD: Undecided
laboratory test